CLINICAL TRIAL: NCT05788107
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of HLX51 (Anti-OX40 Monoclonal Antibody) in Patients With Advanced/Metastatic Solid Tumor or Lymphoma
Brief Title: Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of HLX51 in Patients With Solid Tumor or Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX51-FIH101
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor, Adult Lymphoma
Keywords: OX40
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX51 Group (Experimental): The initial dose of HLX51 is 0.3mg/kg, and 5 dose levels are designed: 0.3 mg/kg, 1 mg/kg , 2.5mg/kg, 5mg/kg, and 10mg/kg (Q3W). Patients with good tolerability and well controlled disease will receive the treatment until progressive disease (PD) without any clinical benefit, initiation of other anti-tumor therapies, death, intolerable toxicity, or withdraw the informed consent (whichever occurs first).
  Interventions: Drug: HLX51

INTERVENTIONS:
Drug: HLX51 — anti-OX40 tetravalent agonistic humanized monoclonal antibody
  Other Names: anti-OX40 monoclonal antibody

SUMMARY:
This study is a first-in-class open-label phase I human clinical study to evaluate the safety and tolerability of HLX51 with escalated doses in the treatment of patients with advanced/metastatic solid tumors or lymphomas.

DETAILED DESCRIPTION:
This study is the first-in-class open-label phase I human clinical study to evaluate the safety and tolerability of HLX51 with escalated doses in the treatment of patients with advanced/metastatic solid tumors or lymphomas. In this study, 3 + 3 dose escalation method will be adopted, and the patients will be given different doses of HLX51 intravenously. Observation period of DLT lasts for 3 weeks after the first administration of HLX51.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF). voluntarily participate in the study. be able to complete the study as per protocol requirements.
2. Aged ≥ 18 years at the time of signing the ICF.
3. Patients with histologically or cytologically confirmed advanced malignant solid tumor or lymphoma, who have failed or cannot receive the standard treatment.
4. With at least one measurable lesion according to RECIST V1.1 (for solid tumors) or the Lugano criteria (for lymphomas).
5. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1 at enrollment.
6. Expected survival > 3 months.
7. Have appropriate hematological functions: no blood transfusion or colony stimulating factor therapy (G-CSF) within 14 days before the first administration. absolute neutrophil count ≥ 1500/μL. haemoglobin ≥ 9 g/dL. platelet count ≥ 90,000/μL.
8. Have appropriate coagulation functions: activated partial thromboplastin time (APTT) ≤ 1.5 × ULN. prothrombin time (PT) ≤ 1.5 × ULN. international normalized ratio (INR) ≤ 1.5 × ULN.
9. Have appropriate liver functions: total bilirubin level ≤ 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN (AST and ALT ≤ 5 × ULN for patients with known liver metastasis or primary hepatocellular carcinoma).
10. Have appropriate renal functions: blood creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula).
11. The first administration of the investigational product must be: at least 28 days apart from the previous major surgery, medical device treatment, or local radiotherapy. at least 28 days apart from the previous cytotoxic chemotherapy, immunotherapy, and biological agent therapy. at least 14 days apart from the previous hormone therapy and surgical operation. at least 21 days or 5 half-lives apart from the administration of small molecule targeted drugs, whichever is longer. at least 14 days apart from the traditional Chinese medicine for tumor indications.
12. For patients with hepatocellular carcinoma, Child-Pugh score has to be A.
13. Male and female subjects with child-bearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months after the last administration of the investigational product.

Exclusion Criteria:

1. Previous exposure to any anti-OX40 antibody or any drug targeting T-cell costimulatory signaling pathway.
2. The adverse reactions (except alopecia and other adverse reactions determined by the investigator to have no safety risk) of previous anti-tumor therapy have not yet recovered to ≤ grade 1 (CTCAE V5.0).
3. Those who are known to have severe anaphylaxis to macromolecular protein preparations/monoclonal antibodies or to any component of the investigational product.
4. Patients with any of the following unstable or poorly controlled diseases:

1) Active systemic infectious diseases requiring intravenous antibiotics within 2 weeks before the first administration of the investigational product.

2) Any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or greater cardiac failure or left ventricular ejection fraction (LVEF) < 50%. (2) unstable angina pectoris. (3) myocardial infarction and cerebral infarction within 6 months, (4) clinically significant supraventricular or ventricular arrhythmia without clinical intervention or poorly controlled after clinical intervention.

3) Other chronic diseases which, in the opinion of the investigator, may compromise the safety of the patient or the integrity of the study.

5. Assessed as unsuitable for inclusion by the investigator, due to brain metastases, spinal cord compression, or cancerous meningitis with clinical symptoms, or uncontrolled brain or spinal cord metastases that have been evidenced.

6. Previous grade 3 or greater irAEs in immunotherapy. 7. Have had other malignant tumors within 5 years before enrollment, except: (a) those with cured cervical carcinoma in situ or non-melanoma skin cancer. (b) those with cured second primary cancer without recurrence within 5 years. (c) those with double primary cancers believed to be able to benefit from this study. (d) those whose metastasis has been clearly excluded from a certain primary tumor source.

8. Have active autoimmune diseases (including but not limited to the following diseases or syndromes, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism), except: vitiligo or cured childhood asthma/allergy that does not need any intervention in adulthood, autoimmune mediated hypothyroidism treated with stable dose of thyroid replacement hormone, and type I diabetes treated with stable dose of insulin. those in a stable condition and requiring no systemic immunosuppressant therapy (including corticosteroid hormone) are allowed to be enrolled.

9. Have received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 14 days before the first administration.

Except: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids. those with short term use of corticosteroids for prophylaxis, such as contrast agents.

10. Patients in pregnancy [confirmed by serum beta-human chorionic gonadotropin (ß-HCG) test] or breastfeeding.

11. With a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or a history of organ transplantation.

12. With a history of interstitial lung disease or active tuberculosis. 13. Patients with active HBV or HCV infection (HBV DNA ≥ 104 copies/mL or positive HCV RNA).

14. Have received live vaccines within 30 days prior to the first administration.

Patients whose medical history or any other evidence suggests that participation in the study may confuse the results, or subjects for whom the investigator believes the study is not in their best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) of HLX51 within 3 weeks after the first Administration | At the end of Cycle 1 (each cycle is 21 days)
  DLT refers to the AEs that are determined to be related to the investigational product by the investigator, whose severity will affect the escalation of dose level. In this study, the DLT observation period lasts for 3 weeks after the first administration of HLX51
The maximum tolerated dose (MTD) of HLX51 within 3 weeks after the first administration | At the end of Cycle 1 (each cycle is 21 days)
  MTD refers to the highest dose at which less than 1/3 of subjects in the same dose group develop DLT in cycle 1 of the dose escalation stage.